CLINICAL TRIAL: NCT02804607
Title: Children Severe Traumatic Skin Lesions and Functional Outcome
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0019
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Burns
Keywords: burn; child; graft; development; complications; autonomy
MeSH Terms: conditions — Burns | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- skin lesion: severe skin traumatism occurring during childhood and which had required an initial graft.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire

SUMMARY:
Traumatic skin lesions require an adapted and early patient care management

DETAILED DESCRIPTION:
Traumatic skin lesions and in particular the burns which happen to growing children are complex and require an adapted and early patient care management. A child presents physical, psychological, and physiological characteristics which involve a specific functional prognosis. The aim of the study was to evaluate the functional outcome after a mid-term period from a severe skin traumatism occurring during childhood and which had required an initial graft.

ELIGIBILITY:
Inclusion Criteria:

* children who were hospitalized for an extensive and deep skin lesion on at least one joint, at CHU Amiens, from April 1999 to December 2014, in the Physical and Rehabilitation Pediatric activity center.
* And with a serious skin lesion:

  * What the total dermal area is estimated to be less than 25%
  * Taking at least one articulation
  * Dont a part is at least 2nd degree deep or third degree

Exclusion Criteria:

* First degree burns or superficial second degree Burns resulting in death in the acute phase
* A history of pre-burn disorders affecting growth
* Escarres

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children who were hospitalized for an extensive and deep skin lesion on at least one joint, at CHU Amiens, from April 1999 to December 2014, in the Physical and Rehabilitation Pediatric activity center.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2016-02-08 (Actual)

PRIMARY OUTCOMES:
autonomy | 5 years
  for daily life activities (questionnaire)

SECONDARY OUTCOMES:
appearance of contractures | 5 years
  consultation follow-up
limited joint mobility | 5 years
  consultation follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Séverine FRITOT, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France